CLINICAL TRIAL: NCT01371578
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Response Guided Therapy Using Combinations of Oral Antivirals (GS-5885, Tegobuvir, and/or GS-9451) With Peginterferon Alfa 2a and Ribavirin in Treatment Experienced Subjects With Chronic Genotype 1 Hepatitis C Virus Infection (Protocol GS US 256 0124)
Brief Title: Oral Antivirals (GS-5885, Tegobuvir, and/or GS-9451) With Peginterferon Alfa 2a and Ribavirin in Treatment Experienced Subjects With Chronic Genotype 1 Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-256-0124
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C; HCV; Rapid Virologic Response; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy HCV RNA; Polymerase inhibitor; Protease inhibitor; Treatment naïve; GS-5885; GS-9190; Tegobuvir; GS-9451
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ledipasvir; GS-9451; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm 2 (Experimental): AM Dosing: One GS-5885 30 mg tablet, two GS-9451 100 mg tablets, orally with RBV and with food.
  PM Dosing: RBV with food.
  PEG, 180 µg, will be administered weekly by subcutaneous injection for the specified period of time (see Study Design). Pegasys® prefilled syringes (Hoffman-La Roche) will be supplied by Gilead Sciences.
  Interventions: Drug: GS-5885 tablet; Drug: GS-9451 tablet; Biological: peginterferon alfa-2a; Drug: ribavirin tablet

INTERVENTIONS:
Drug: GS-5885 tablet — 30 mg active tablet
Drug: GS-9451 tablet — two active 100 mg tablets
Biological: peginterferon alfa-2a — peginterferon alfa-2a (solution for injection) 180 µg/week
Drug: ribavirin tablet — ribavirin tablet (weight based: 1000 mg/day <75 kg; 1200 mg/day ≥ 75 kg) divided twice daily (BID); tablet

SUMMARY:
This is a Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial Evaluating Response Guided Therapy using Combinations of Oral Antivirals (GS-5885, tegobuvir, and/or GS-9451) with Peginterferon Alfa 2a and Ribavirin in Treatment Experienced Subjects with Chronic Genotype 1 Hepatitis C Virus (HCV) Infection.

DETAILED DESCRIPTION:
In September 2011, the FDA requested that Gilead make several major changes to this study because of side effects experienced by two patients in other Gilead studies.

In 2 HCV-infected people that were given tegobuvir with another experimental medication plus interferon and ribavirin, big reductions in the number of white blood cells, red blood cells and platelets were seen. Because these cases might have been related to tegobuvir when given with interferon, ribavirin and another direct antiviral agent, tegobuvir is no longer being given to people with these other medications in this study.

As a result, the study is now open label which means both you and your study doctor will know the medication you will be receiving and Arms 1 and 3 have been discontinued from the study.

All subjects enrolled in the study as of September 2nd 2011 will receive Response Guided Therapy (RGT) with both GS-5885 and GS-9451 plus PEG and RBV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18 to 70 years old, inclusive
* Chronic HCV infection for at least 6 months prior to Baseline
* Subjects must have liver biopsy results (≤ 3 years prior to screening) indicating the absence of cirrhosis.
* Monoinfection with HCV genotype 1
* HCV RNA > 10^4 IU/mL at Screening
* Prior treatment and adherence (as defined by receiving at least 80% of the prescribed treatment) with one course of a pegylated interferon-alfa (Pegasys or Peg-Intron) and RBV
* The subject's medical records must include sufficient detail of prior treatment with pegylated interferon-alfa and RBV (start/stop dates and viral response) to allow for categorization of prior response as either

  * Non-Responder: Subject did not achieve undetectable HCV RNA levels during or at the end of a treatment period of at least 12 weeks duration. Within Nonresponders, subjects will be further defined as Null or Partial Responders if they had < 2 log10 or ≥ 2 log10 reduction, respectively, in HCV RNA during the first 12 weeks of treatment
  * Responder: Subject achieved undetectable HCV RNA during treatment. Within Responders, subjects will be further defined as Relapsers if they had undetectable HCV RNA at the end of at least 42 weeks of treatment but detectable HCV RNA levels observed within 1 year of the end of treatment and Breakthrough subjects if they achieved undetectable HCV RNA levels during the treatment period but detectable HCV RNA at the end of treatment.
* No prior treatment with an oral HCV antiviral (exclusive of RBV).
* Body mass index (BMI) 18-36 kg/m2, inclusive.
* Screening ECG without clinically significant abnormalities and with QTcF interval (QT corrected using Fridericia's formula) ≤ 450 msec for males and ≤ 470 msec for females
* Creatinine clearance ≥ 50 mL/min.
* Agree to use two forms of highly effective contraception for the duration of the study and for 6 months after the last dose of study medication. Females of childbearing potential must have a negative pregnancy test at Screening and Baseline

Exclusion Criteria:

* Discontinued prior treatment with pegylated interferon-alfa and RBV due to an adverse event, toxicity reasons or were lost to follow-up.
* Exceed defined thresholds for leukopenia, neutropenia, anemia, thrombocytopenia, thyroid stimulating hormone (TSH)
* Diagnosis of autoimmune disease, decompensated liver disease, poorly controlled diabetes mellitus, significant psychiatric illness, severe chronic obstructive pulmonary disease (COPD), HIV, hepatitis B virus (HBV), or another HCV genotype, hepatocellular carcinoma or other malignancy (with exception of certain skin cancers), hemoglobinopathy, retinal disease, or are immunosuppressed.
* Current use of amphetamines, cocaine, opiates (e.g., morphine, heroin), or ongoing alcohol abuse are excluded. Subjects on stable methadone are excluded, however stable buprenorphine maintenance treatment for at least 6 months is not exclusionary
* Receiving any of the prohibited concomitant medications.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) | through 24 weeks of off-treatment follow-up
  To evaluate antiviral efficacy as measured by sustained virologic response (SVR, defined as HCV RNA < Lower Limit of Quantification (LLoQ) 24 weeks post-treatment) of response guided therapy (RGT) with GS-9451 + GS-5885, with peginterferon alfa-2a (PEG) and ribavirin (RBV) in treatment-experienced subjects.

SECONDARY OUTCOMES:
Sustained Virologic Response(SVR) of each regimen administered for 24 to 48 weeks | Weeks 1, 2, 4, 8, 12, 16, 20, 24, 36, 48 and at 4 and 12 weeks off-treatment
  To evaluate antiviral efficacy as measured by SVR for 24 or 48 weeks of treatment with GS-5885, GS-9451, PEG, RBV.
Safety and Tolerability | through 24 to 48 week treatment period and up to 24 weeks of off-treatment follow-up
  To evaluate the safety and tolerability of treatment with GS-5885, GS-9451, PEG & RBV administered for 24 or 48 weeks. Safety endpoints will be summarized as the number (proportion) of subjects with events or abnormalities for categorical values or as an 8-number summary (n, mean, standard deviation, median, Q1, Q3, minimum, maximum) for continuous data by treatment arm.
Characterize the viral dynamics of GS-5885, GS-9451 when administered in combination with PEG and RBV | Through Week 2 of therapy
  HCV RNA levels, pharmacokinetics, and viral sequencing
Characterize the pharmacokinetics of GS-5885 and GS-9451 when administered in combination with PEG and RBV | Through Week 2 of therapy
  Plasma concentrations of the study drug over time will be summarized using descriptive statistics. Pharmacokinetic parameters (Cmax, Tmax, Clast, Tlast, Ctau, λz, AUCtau, and T½) will be listed and summarized for GS-5885 and GS-9451, using descriptive statistics (eg, sample size, arithmetic mean, geometric mean, % coefficient of variation, standard deviation, median, minimum, and maximum).
Emergence of Viral Resistance | through 24 to 48 week treatment period and up to 24 weeks of off-treatment follow-up
  To characterize the viral resistance to GS-5885 and GS 9451tegobuvir when administered in combination with PEG and RBV.

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Chair — Gilead Sciences
Locations (55):
- United States (54):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Alabama Liver and Digestive Specialists, Montgomery, Alabama
  - California Liver Institute, Beverly Hills, California
  - Scripps Clinic, La Jolla, California
  - University of California Davis Medical Center, Sacramento, California
  - RESEARCH and EDUCATION, INC, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - Kaiser Permanente, San Diego, California
  - University of Colorado Denver, Aurora, Colorado
  - South Denver Gastroenterology, Englewood, Colorado
  - Bach and Godofsky Infectious Diseases, Bradenton, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - South Florida Center of Gastroenterology, LLC, Wellington, Florida
  - Emory University, Infectious Disease Clinic, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Dekalb Gastroenterology, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Digestive Disease Associates, PA, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Partners in Internal Medicine, P.C., Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - ID Care 105, Hillsborough, New Jersey
  - Atlantic Research Affiliates, LLC, Morristown, New Jersey
  - Southwest CARE Center, Santa Fe, New Mexico
  - Binghamton Gastroenterology, Binghamton, New York
  - North Shore University Hospital, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - Cornell University Gastroenterology & Hepatology, New York, New York
  - Asheville Gastroenterology Associates, P.A., Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Options Health Research, LLC, Tulsa, Oklahoma
  - University Gastroenterology, Providence, Rhode Island
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Columbia Medical Group, The Frist Clinic, Nashville, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Nashville Gastrointestinal Specialists, Inc, Nashville, Tennessee
  - The North Texas Research Institute, Arlington, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Research Specialists of Texas, Houston, Texas
  - Metropolitan Research, Fairfax, Virginia
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - Liver Institute of Virginia, Richmond, Virginia
  - Virginia Mason Medical Center, Digestive Disease Institute, Seattle, Washington
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico